CLINICAL TRIAL: NCT03546933
Title: A Prospective Multi-centre Observational Study to Validate the Diagnostic Accuracy of a Transportable Magnetocardiograph Device for Acute Coronary Syndrome (ACS), Focusing on Rule-out Capability, in Patients Who Present to the Emergency Department With Chest Pain Symptoms Consistent With ACS
Brief Title: VitalScan MCG Rule-out Multi-centre Pivotal Study - US
Acronym: MAGNET ACS
Status: Terminated | Type: Observational
Why Stopped: A correction needs to be made to the device's algorithm.
Sponsor: Creavo Medical Technologies Ltd (Industry)
Collaborators: University of Cincinnati (Other)
Responsible Party: Sponsor
Other Study IDs: CIP 003 (US)
Record Dates: First submitted 2018-05-09; First posted 2018-06-06 (Actual); Last update posted 2019-09-18 (Actual); Status verified 2019-09

CONDITIONS: Acute Coronary Syndrome
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Chest pain patients presenting to the ED: All patients that present to the emergency department with chest pain and potentially other symptoms consistent with ACS and meet all eligibility criteria will undergo VitalScan Magnetocardiograph.
  Interventions: Device: VitalScan Magnetocardiograph

INTERVENTIONS:
Device: VitalScan Magnetocardiograph — A passive, non-contact, mobile medical device that measures, displays, stores, and retrieves magnetic fluctuations caused by heart activity at a patient's bedside.

SUMMARY:
A prospective multi-centre observational study to validate the diagnostic accuracy of a transportable magnetocardiograph device for acute coronary syndrome (ACS), focusing on rule-out capability, in patients who present to the emergency department with chest pain symptoms consistent with ACS.

ELIGIBILITY:
Inclusion Criteria:

* Patient presents to the ED with chest pain syndrome of suspected cardiac origin (i.e. symptoms consistent with ACS)
* 18+ year old male or female
* Patient is willing and able to give written informed consent

Exclusion Criteria:

* ST-segment Elevation MI (STEMI)
* Clear non-ischemic cause for symptoms (e.g. trauma)
* Hemodynamic instability on admission (e.g. BP>220mmHg systolic & >110mmHg diastolic, <80mmHg systolic & <40mmHg diastolic, HR>160bpm)
* Ventricular tachycardia or fibrillation that cannot be treated effectively
* Atrial fibrillation
* Thoracic metal implants
* Pacemaker or internal defibrillator
* Pregnancy (if after 20-week period)* or lactation
* Patient unable to lie down (i.e. supine position) or stay still on the examination bed
* Patient unable to understand the informed consent process and/or has a poor understanding of English (e.g. English- speaking relative/translator not available)
* Patient unable to comply with the requirements of the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients that present to the ED with chest pain syndrome of suspected cardiac origin (i.e. symptoms consistent with ACS) who are in normal sinus rhythm
Sampling Method: Probability Sample
Enrollment: 651 (Actual)
Dates: Start 2018-07-17 (Actual); Primary Completion 2019-08-06 (Actual); Study Completion 2019-08-06 (Actual)

PRIMARY OUTCOMES:
Sensitivity and specificity of MCG | up to 3 month follow-up
  Sensitivity and specificity for diagnosing ACS, focusing on rule-out, in chest pain patients with normal sinus rhythm

SECONDARY OUTCOMES:
Proportion of adverse events and types | up to 3 month follow-up
All-cause mortatility (divided into CV and non-CV causes) proportion | through 1 week, 3 month follow-up
3.Change in sensitivity and specificity for diagnosing ACS, focusing on rule-out, in chest pain patients with normal sinus rhythm, according to low, intermediate and high PTP groups | up to 3 months follow-up
MACE post-presentation to the ED (rule-out of ACS divided into MCG vs reference standard (adjudicated ACS/non-ACS diagnoses)) | through 1 week, 3 month follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Gregory J Fermann, MD, Principal Investigator — University of Cincinnati
Locations (5):
- United States (5):
  - IU Health Methodist Hospital, Indianapolis, Indiana
  - Wake Forest Baptist Medical Center, Winston-Salem, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Baylor College of Medicine, Houston, Texas

IPD SHARING:
Plan to Share IPD: No